CLINICAL TRIAL: NCT00928213
Title: Combined Sonographic Examination and Placenta Protein 13 (PP13) to Compare the Risk for Development of Preeclampsia Among Among Pregnant Women With and Without a History of Preterm Delivery and Those Treated by Progesterone or Clexane
Brief Title: PP13 and Doppler Study to Predict Preeclampsia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ben-Gurion University of the Negev (Other)
Collaborators: Diagnostic Technologies Ltd. (Industry); Perkin Elmer Inc. (Industry); Medical University of Graz (Other)
Responsible Party: Dr. Reli Hershkovitz, Soroka Medical Center Ben Gurion University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 972-07-024
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2009-06

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; IUGR; GH; PP13; Doppler; placenta; PTD; Preterm delivery
MeSH Terms: conditions — Pre-Eclampsia; Premature Birth | interventions — Progesterone; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Control not treated, no placebo
  Interventions: Drug: No Drug
- 2 (Experimental): Patient treated with low molecular weight heparin after repeated pregnancy loss
  Interventions: Drug: Low molecular weight Heparin
- 3 (Experimental): Patient super from first trimester bleeding treated with progesterone
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — 40 units daily admission
  Other Names: C-21 steroid hormone; Prometrium
  Arms: 3
Drug: Low molecular weight Heparin — 40-80 mg/day
  Other Names: clexan
  Arms: 2
Drug: No Drug — no treatment
  Other Names: No treatment
  Arms: 1

SUMMARY:
Assessment of biochemical and sonographic marker to predict the risk for developing preeclampsia Among biochemical markers are serum level of Placental Protein 13 (PP13) and Placenta Growth factor (PIGF). For sonographic marker Doppler pulsatility Index of the blood flow through the uterine maternal arteries is assessed.

PP13 is produced by the placenta and released to the maternal blood circulation. It has been shown to be an effective serum marker for early onset preeclampsia (Nicolaides KH et al., 2005). The purpose of this study is to combined the assessment of the biochemical markers with Doppler in the first and the second trimester to provide a comprehensive evaluation of various methods for sequential and combined analysis to assess the risk for developing preeclampsia.

DETAILED DESCRIPTION:
This is a prospective observational study enrolling all comers who attend the prenatal clinic for first trimester assessment of the risk for Down syndrome. All women are providing medical and obstetric history, demography and blood samples along with Doppler pulsatility Index during the first and the second trimester at GA 10-13 weeks and 21-23 weeks. When possible - blood will be drawn at hospital admission for delivery. Measurements of sonography and serum markers are done blinded to pregnancy outcome.

Patients will be assigned to three groups:

1. All comers attending the prenatal testing at GA 10-13.
2. Patients with a history of at least 2 pregnancy loss or preterm delivery and treated with low molecular weight heparin at 40-80 mg/day from admission to until 12 weeks after delivery.
3. Patients who admitted the emergency ObGyn clinic for bleeding during the first trimester and are treated with progesterone.

ELIGIBILITY:
Inclusion Criteria:

* Women age 16-45 with viable pregnancy as defined by CRL and after signing on an informed consent
* In group 1 all patients meeting the above are eligible when GA is below 14 weeks
* In grop 2 all patients

Exclusion Criteria:

* Gestation age at enrolment > 13 weeks and 6 days by LMP verified by ultrasound at blood taking
* Mental retardation or other mental disorders that impose doubts regarding the patient's true willingness to participate in the Study

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Preeclampsia (hypertension >140/90, proteinuria >2+ or 300 mg/Dl in 24 hr collection | pregnancy week >20 till 41 weeks

SECONDARY OUTCOMES:
intra uterine growth restriction, preterm delivery, spontaneous abortion and Intra uterine fetal death | fron conception to until a week after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Reli Hershkovitz, MD, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Soroka Medical Center, Ben Gurion University, Beersheba, Israel

REFERENCES:
- See also: The website of Ben Gurion University — http://www.bgu.ac.il